CLINICAL TRIAL: NCT03198013
Title: Placebo-Controlled, Double-Blind, Ascending Single and Multiple Oral Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-791826 and to Assess Its Marker Specific Pharmacodynamics in Relation to Prednisolone in Healthy Males
Brief Title: A Study of Pharmacokinetics (PK) and Pharmacodynamics (PD) in Relation to Prednisolone in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IM125-001
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Immunoscience
MeSH Terms: interventions — Prednisolone; 5-2-(4-((ethylmethylamino)carbonyl)-3-fluorophenyl)-alpha,alpha-dimethyl-N-1,3,4-thiadiazol-2-yl-5H-(1)benzopyrano(2,3-b)pyridin-5-acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Module A (Experimental): Single Ascending Dose
  Interventions: Drug: Prednisolone; Drug: BMS-791826; Drug: Placebo
- Module B (Experimental): Multiple Ascending Dose
  Interventions: Drug: Prednisolone; Drug: BMS-791826; Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — Specified dose on specified days
Drug: BMS-791826 — Specified dose on specified days
Drug: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, PK, PD, of BMS-791826 and to assess its marker specific PD in relation to Prednisolone in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 30 kilogram / square meter (kg/m2), inclusive
* Signed informed consent

Exclusion Criteria:

* Sexually active fertile men not using effective birth control (barrier contraception) if their partners are women of childbearing potential (WOCBP)
* Any significant acute or chronic medical illness
* History of Gilbert's disease

Other protocol inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11-11 (Actual); Primary Completion 2009-05-18 (Actual); Study Completion 2009-05-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 34 days
  safety and tolerability
Incidence of serious adverse events (SAEs) | Up to 34 days
  safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Hu Y, Carman JA, Holloway D, Kansal S, Fan L, Goldstine C, Lee D, Somerville JE, Latek R, Townsend R, Johnsen A, Connolly S, Bandyopadhyay S, Shadick N, Weinblatt ME, Furie R, Nadler SG. Development of a Molecular Signature to Monitor Pharmacodynamic Responses Mediated by In Vivo Administration of Glucocorticoids. Arthritis Rheumatol. 2018 Aug;70(8):1331-1342. doi: 10.1002/art.40476. Epub 2018 Jul 12. PMID 29534336